CLINICAL TRIAL: NCT03094533
Title: The Effect of Total Intravenous Anesthesia and Volatile Induction and Maintenance Anesthesia on Perioperative Blood Glucose and Insulin Levels in Patients Undergoing Lung Lobectomy
Brief Title: TIVA and VIMA on Blood Glucose and Insulin Levels in Lung Lobectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sung Mee Jung, Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YUMC 2017-02-036
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Hyperglycemia Stress
Keywords: Anesthesia, intravenous; Anesthesia, inhalation; propofol; sevoflurane; glucose
MeSH Terms: conditions — Respiratory Aspiration | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total intravenous anesthesia (Active Comparator): In the total intravenous anesthesia(TIVA) group, target controlled infusion (TCI) I was performed with propofol 4 mcg / ml. When the consciousness of the patient is lost, Remifentanil is administered as TCI with a target concentration of 1 ng / ml as an analgesic agent, and rocuronium 0.5 mg / kg is administered intravenously for intubation.
  Interventions: Drug: TIVA
- volatileinduction maintenance anesthesia (Active Comparator): In the volatile induction and maintenance anesthesia(VIMA) group, when 8% sevoflurane is inhaled with 100% oxygen at 6 L / min and the consciousness is lost, the concentration of sevoflurane is reduced to 2-3% and then the mask is ventilated.Remifentanil is administered as TCI with a target concentration of 1 ng / ml as an analgesic agent, and rocuronium 0.5 mg / kg is administered intravenously for intubation.
  Interventions: Drug: VIMA

INTERVENTIONS:
Drug: TIVA — total intravenous anesthesia with propofol
  Other Names: propofol
  Arms: Total intravenous anesthesia
Drug: VIMA — volatile induction and maintenance anesthesia with sevoflurane
  Other Names: sevoflurane
  Arms: volatileinduction maintenance anesthesia

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of sevoflurane-only Volatile induction and maintenance anesthesia (VIMA) and total intravenous anesthesia (TIVA) using only propofol in adult patients scheduled for elective lobectomy surgery. We would like to know if there is a difference in blood glucose levels during surgery and whether the cause is due to the difference in secretion of insulin and cortisol. In addition, we aim to contribute to the improvement of the prognosis of the patients by helping the selection of general anesthesia more effective in maintaining homeostasis in the surgical patients by general anesthesia and further controlling the blood glucose level.

DETAILED DESCRIPTION:
Before surgery, glycopyrrolate (0.2 mg) was administered intramuscularly. Immediately after arrival in the operating room, blood pressure, electrocardiogram and oxygen saturation are measured and monitored, and a bispectral index (BIS) is attached to the patient's forehead to determine the appropriate anesthetic depth during surgery. A 22G angiocatheter is inserted into the radial artery after local anesthesia with lidocaine to monitor the blood pressure in real time and to collect blood for arterial blood gas analysis during one side of pulmonary ventilation. General anesthesia induces loss of consciousness by using a randomly assigned systemic anesthetic (sevoflurane inhalation or propofol infusion). In the VIMA group, when 8% sevoflurane is inhaled with 100% oxygen at 6 L / min and the consciousness is lost, the concentration of sevoflurane is reduced to 2-3% and then the mask is ventilated. In the TIVA group, target controlled infusion (TCI) was performed with propofol 4 mcg / ml, and the patient was ventilated after disappearance of consciousness. When the consciousness of the subject is lost, remifentanil is administered as TCI with a target concentration of 1 ng / ml as an analgesic agent, and rocuronium 0.5 mg / kg is administered intravenously for intubation in both groups. If the patient's anesthesia depth is between BIS 40-60 and the respiratory muscles are fully relaxed, tracheal intubation is performed using the double lumen endobronchial tube (DLT). After confirming the DLT reaches the proper position with a flexible bronchoscope, mechanical ventilation is started by administering 50% oxygen. The central venous catheter is inserted into the operative subclavian vein and the central venous pressure is continuously monitored during the operation. During surgery, rocuronium is administered continuously so that the train-of-four (TOF) remains below two responses. In addition, warm blanket and warm air are supplied to the rest of the body except for the surgical site so that the patient can maintain normothermia during the operation. In all patients, surgery should start between 8:30 am and 9:00 am in order to prevent volatility of blood cortisol levels by activity cycle. During surgery, general anesthesia should be adjusted to maintain BIS 40-60, and remifentanil TCI should be maintained at 1 ng / ml for pain during surgery. The mean blood pressure during surgery is aimed at maintaining a 30% range on baseline so that hypotension or hypertension does not last more than 5 minutes. Hypotension and hypertension are controlled by intravenous injection of phenylephrine (50 μg / ml) and nicardipine (500 μg / ml), respectively. At the end of the operation and after the paravertebral block to control the postoperative pain, the administration of the general anesthetic and remifentanil is stopped and the spontaneous breathing is tried to be recovered. When patients begin spontaneous breathing, the effect of the remaining neuromuscular blockers is reversed using pyridostigmine (0.2 mg / kg) and glycopyrrolate (0.008 mg / kg). All patients are fully conscious and have a spontaneous respiration when they are exhaled and transferred to the postanesthetic care unit (PACU). PACU administers oxygen through a facial mask and monitors blood pressure, heart rate and oxygen saturation. Patients should be given 1 ug / kg of fentanyl when the visual analog scale (VAS) scores exceed 4 points

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic patients American Society of Anesthesiologist Physical Status Classification 1 - 3

Exclusion Criteria:

* Diabetes mellitus or glucose intolerance patients, patients with adrenocortical hormone metabolism abnormality, patients with steroids therapy within the last month, patients with liver disease (aspartate aminotransferase> 40 IU / L or alanine aminotransferase> 40 IU / L), patients with kidney disease (creatinine 1.5 mg / dl), pregnant woman, patients with hypersensitivity to anesthetics used in research, patients who required ventilator care after surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Perioperative glucose level | up to 1 hour after surgery
  The blood glucose level measured by the patient's blood sample

SECONDARY OUTCOMES:
Perioperative insulin and cortisol levels | Baseline, 1 hour after incision, intraoperative, 1 hour after surgery
  Insulin and cortisol concentrations measured in blood samples of patient

CONTACTS AND LOCATIONS:
Overall Officials: Sung Mee Jung, MD,PhD, Principal Investigator — Yeungnam University Hospital
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Cok OY, Ozkose Z, Pasaoglu H, Yardim S. Glucose response during craniotomy: propofol-remifentanil versus isoflurane-remifentanil. Minerva Anestesiol. 2011 Dec;77(12):1141-8. Epub 2011 May 20. PMID 21602751
- [Result] Kitamura T, Kawamura G, Ogawa M, Yamada Y. [Comparison of the changes in blood glucose levels during anesthetic management using sevoflurane and propofol]. Masui. 2009 Jan;58(1):81-4. Japanese. PMID 19175019
- See also: Isoflurane and propofol, both combined with remifentanil, provided clinically comparable cortisol and insulin responses to surgery in craniotomy operations, whereas propofol attenuated the increase in plasma blood glucose — https://www.ncbi.nlm.nih.gov/pubmed/?term=OY+Cok%2C+Z+Ozkose%2C+H+Pasaoglu%2C+S+Yardim+%3A+Glucose+response+during+craniotomy%3A+propofol
- See also: Results in this study imply that the effect on glucose metabolism of propofol is much less than that of sevoflurane — https://www.ncbi.nlm.nih.gov/pubmed/?term=Kitamura+T%2C+Kawamura+G%2C+Ogawa+M%2C+Yamada+Y+%3A+Comparison+of+the+changes+in+blood